CLINICAL TRIAL: NCT01671839
Title: Pivotal Study of the Cabochon System for Improvement in the Appearance of Cellulite
Brief Title: Study of the Cabochon System for Improvement in the Appearance of Cellulite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Collaborators: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-01-1004
Record Dates: First submitted 2012-08-17; First posted 2012-08-24 (Estimated); Results first posted 2014-09-04 (Estimated); Last update posted 2019-12-10 (Actual); Status verified 2019-08

CONDITIONS: Gynoid Lipodystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Subcutaneous tissue release (Experimental): Device: Subcutaneous tissue release with the Cabochon System
  Interventions: Device: Subcutaneous tissue release with the Cabochon System

INTERVENTIONS:
Device: Subcutaneous tissue release with the Cabochon System — Device: Subcutaneous tissue release
  Other Names: Cellfina®

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Cabochon System for the improvement in the appearance of cellulite.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18-55
* moderate or severe cellulite
* BMI less than 35
* will not to try any other cellulite treatments through 12M follow-up

Exclusion Criteria:

* cellulite treatment on the thighs or buttocks in the last 90 days
* prior liposuction in the thighs or buttocks
* Greater than 10% increase or decrease in body weight within past 6 months
* evidence of active infection or a fever >38C
* current or recent smoker
* history of hypertension, diabetes or hypoglycemia
* history of coagulopathy(ies) and/or on anticoagulant medication
* history of cardiopathy or pneumopathy
* history of severe anemia
* has atrophic scars, or has a history of atrophic scars or keloids
* taken within 14 days of treatment:

  * NSAIDs (e.g. aspirin, ibuprofen, naproxen)
  * Vitamin E, dietary supplements (e.g. Gingko Biloba, willow bark)
  * Herbal Teas
* Subject is pregnant or lactating

For Extended Follow-Up the following apply:

Inclusion Criteria:

* Subject was enrolled and treated in the CP-01-1004 study - Pivotal Study of the Cabochon System for Improvement in the Appearance of Cellulite
* Subject understands and accepts the obligation not to try or receive any other cellulite treatments through 3 year follow-up

Exclusion Criteria:

* Subject has undergone an injected drug, energy-based device, minimally-invasive or invasive procedure for contouring or cellulite on the buttocks or thighs since their 12 month study follow-up visit.
* Subject has used skin care products (e.g. creams) for improvement in cellulite within 1 month prior to the follow-up visit.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2012-08; Primary Completion 2013-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Kaminer, Principal Investigator — Skin Care Physicians
Locations (3):
- United States (3):
  - The Coleman Center for Cosmetic and Dermatologic Surgery, Metairie, Louisiana
  - Maryland Laser Skin & Vein Institute, Hunt Valley, Maryland
  - SkinCare Physicians, Chestnut Hill, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subcutaneous Tissue Release
Started | 55
3-year Follow-up | 45
5-year Follow-up | 37
Completed | 37
Not Completed | 18

BASELINE CHARACTERISTICS:
Arm/Group | Subcutaneous Tissue Release
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.7 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change (Decrease) in Cellulite Severity
Description: Achievement of ≥1 point mean reduction in the 0-5 point Cellulite Severity Scale as determined by independent physician assessment of subject photographs taken before and 3 and 5 years after treatment. Cellulite severity was graded on a 0 (no cellulite) to 5 (severe cellulite) for each subject photograph taken at baseline (before treatment) and 3 and 5 years after treatment by an independent and blinded physician panel. The primary endpoint was achievement of a mean post-treatment severity at 3 and 5 years for the study population which was a minimum of 1 point lower than the baseline severity.
Time Frame: Treatment to 3 and 5 years
Population: The primary analysis was based upon the complete case population (CC). A supportive analysis was generated on the per-protocol (PP). Best-case, worst-case and multiple imputation techniques were utilized to impute missing primary and powered secondary endpoint outcomes.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Subcutaneous Tissue Release
Number analyzed (Participants) | 45
units on a scale
  3 years | 2.0 [1.7 to 2.3]
  5 years: number analyzed (Participants) | 37
  5 years | 1.8 [1.4 to 2.2]

2. Secondary Outcome: Improvement in Cellulite Severity Grade
Description: Percentage of subjects which were scored to have improvement of one grade or more in a 4 point Severity Grade (none, mild, moderate, severe) as determined by independent blinded physician assessment of subject photographs taken before and 3 and 5 years after treatment.
Time Frame: 3 and 5 years
Population: The primary analysis was based upon the complete case population (CC). A supportive analysis was generated on the per-protocol (PP). Best-case, worst-case and multiple imputation techniques were utilized to impute missing endpoint outcomes.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Subcutaneous Tissue Release
Number analyzed (Participants) | 45
percentage of subjects
  3 years | 91.1 [79.3 to 100]
  5 years: number analyzed (Participants) | 37
  5 years | 86 [75 to 100]

3. Secondary Outcome: Improved Appearance
Description: Improvement in subject's cellulite appearance according to a Global Aesthetic Improvement Scale (GAIS) evaluated by independent and blinded physician panel assessment of subject photographs taken before and 3 and 5 years after treatment. Change in the cellulite severity was rated according to 5 measures:
  * Very much improved: Optimal cosmetic result in the treated areas for this subject
  * Much improved: Marked or significant improvement in appearance of the treated areas from the initial condition
  * Improved: Noticeable improvement in appearance of the treated areas from the initial condition but more subtle in magnitude
  * No Change: The appearance of the treated areas is essentially the same as the original condition
  * Worse: The appearance of the treated areas is worse than the original condition
Time Frame: Treatment to 3 and 5 years
Population: The primary analysis was based upon the complete case population (CC).
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Subcutaneous Tissue Release - 3 Years: Device: Subcutaneous tissue release with the Cabochon System
  Subcutaneous tissue release with the Cabochon System: Device: Subcutaneous tissue release
Arm/Group | Subcutaneous Tissue Release - 3 Years | Subcutaneous Tissue Release - 5 Years
Number analyzed (Participants) | 45 | 37
percentage of subjects
  Very Much Improved | 8.9 [2.5 to 21.2] | 5.4 [0.7 to 18.2]
  Much Improved | 46.7 [31.7 to 62.1] | 29.7 [15.9 to 47.0]
  Improved | 44.4 [29.6 to 60] | 64.9 [47.5 to 79.8]
  No Change | 0 [0 to 6.9] | 0 [0 to 9.5]
  Worse | 0 [0 to 6.9] | 0 [0 to 9.5]

4. Secondary Outcome: Subject Satisfaction
Description: Subject rated satisfaction according to a 5 point Likert scale after treatment:
  Very Satisfied Satisfied Neutral Unsatisfied Very Unsatisfied
Time Frame: Treatment to 3 and 5 years
Population: The primary analysis was based upon the complete case population (CC).
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Subcutaneous Tissue Release - 3 Years | Subcutaneous Tissue Release - 5 Years
Number analyzed (Participants) | 45 | 37
percentage of subjects
  % Very Satisfied | 42.2 [27.7 to 57.9] | 46.0 [29.5 to 63.1]
  % Satisfied | 51.1 [35.8 to 66.3] | 32.4 [18.0 to 49.8]
  % Neutral | 6.7 [1.4 to 18.3] | 18.9 [8.0 to 35.2]
  % Unsatisfied | 0 [0 to 6.8] | 0 [0 to 9.5]
  % Very Unsatisfied | 0 [0 to 6.8] | 0 [0 to 9.5]

5. Secondary Outcome: Procedure Tolerability
Description: Subject rated pain according to a 0-10 numerical rating scale. Pain scale ranges from 0 (no pain) to 10 (worst possible pain). Measure was reported as mean and standard deviation of the pain score
Time Frame: Treatment to 3 and 5 years
Population: The primary analysis was based upon the complete case population (CC).
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Subcutaneous Tissue Release - 3 Years | Subcutaneous Tissue Release - 5 Years
Number analyzed (Participants) | 45 | 37
units on scale | 0 (0) | 0 (0)

6. Secondary Outcome: Safe Treatment
Description: Freedom from serious adverse events directly attributable to the Cabochon System or procedure.
Time Frame: Treatment to 3 and 5 years
Measure: Number; unit: occurence of serious adverse events
Arm/Group | Subcutaneous Tissue Release - 3 Years | Subcutaneous Tissue Release - 5 Years
Number analyzed (Participants) | 45 | 37
occurence of serious adverse events | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline up to year 5.
Arm/Group | Subcutaneous Tissue Release - 3 Years | Subcutaneous Tissue Release - Years 4-5
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/37
Other Adverse Events (participants affected / at risk) | 4/55 | 0/37
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Subcutaneous Tissue Release - 3 Years (N=55) | Subcutaneous Tissue Release - Years 4-5 (N=37)
Cold (Infections and infestations) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Hypercholesterolemia (Metabolism and nutrition disorders) | 2 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agrees that the first publication of the results shall be made in conjunction with the results from all study centers. If Investigator desires independently to publish information about data obtained at Investigator's facility, then Investigator may do so, provided a copy of any proposed oral presentation or written publication is received by Company at least 45 days in advance of submission for publication.